CLINICAL TRIAL: NCT07126405
Title: Provider Randomized Trial of the PROvider ReMote ObsTetric-Related Employment Education (PROMOTE)
Brief Title: Provider RCT PROMOTE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been combined with the patient portion of this study under Pro00116081
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00118409; 1R01HD115609-01 (NIH)
Record Dates: First submitted 2025-08-05; First posted 2025-08-17 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Maternal Health; Pregnancy; Employment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving Provider PROMOTE Training (Experimental): Providers in this arm will receive training on PROMOTE
  Interventions: Other: PROvider ReMote ObsTetric-Related Employment Education (PROMOTE)
- Usual Care (No Intervention): Providers in this arm will continue usual care.

INTERVENTIONS:
Other: PROvider ReMote ObsTetric-Related Employment Education (PROMOTE) — An on-demand 30-minute web-based training for clinical team members that provides a high-level summary of federal employment laws, work note templates embedded into the electronic health record (EHR) that prompt the clinician team member to include relevant information, and a patient-facing infographic designed to facilitate clinician counseling.
  Arms: Receiving Provider PROMOTE Training

SUMMARY:
Research Aim 1: Determine the effectiveness of PROMOTE vs. usual care to increase patients' receipt of counseling about workplace accommodations and pregnancy. We will recruit and randomize Obstetric providers to the PROMOTE intervention or usual care. The investigators will compare the frequency of EHR documented work- related counseling and adherence to employer documentation recommendations between the two study arms.

Hypothesis: Patients receiving care by a provider randomized to PROMOTE will have higher rates of documented counseling about work and pregnancy.

Research Aim 2: Determine the effectiveness of PROMOTE vs. usual care to reduce undesired wage or advancement reduction, increase accommodation requests granted, and improve maternal-infant health. The investigators will recruit a racially and socioeconomically diverse cohort of 304 pregnant patients and compare responses to surveys and qualitative interviews about work experiences and EHR-documented maternal-infant health outcomes among patients receiving care by providers randomized to PROMOTE vs. usual care.

Hypothesis: Compared to patients receiving care by providers randomized to usual care, participants receiving care by providers randomized to PROMOTE will have less undesired loss of wages and advancement, increased accommodation request granted, and improved maternal-infant health during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical team member (doctor, nurse, advanced practice provider, any medical assistant or administrative staff)

Exclusion Criteria:

* Not a clinical team member

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of EHR (electronic health record) documented work-related counseling | Up to 1 year
  Used to determine the effectiveness of PROMOTE vs. usual care to increase patients' receipt of counseling about workplace accommodations and pregnancy.
Number of participants who adhere to employer documentation recommendations | Up to 1 year
  Used to determine the effectiveness of PROMOTE vs. usual care to increase patients' receipt of counseling about workplace accommodations and pregnancy.
Number of participants with undesired wage or advancement reduction | Up to 1 year
  Determined by responses to surveys and qualitative interviews about work experiences.
Number of participants with accommodation requests granted | Up to 1 year
  Determined by responses to surveys and qualitative interviews about work experiences.
Number of participants with improved maternal-infant health in pregnancy | Up to 1 year
  Determined by EHR-documented maternal infant health outcomes among patients receiving care by providers randomized to PROMOTE vs. usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Sarahn Wheeler, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No